CLINICAL TRIAL: NCT02424409
Title: Evaluation of the Relapse Rate One Month After Discharge From Emergency Department for Asthmatic Patients Given a Strict Formalized Follow up Protocol. Multicenter, Prospective, Cluster-randomized
Brief Title: Evaluation of the Relapse Rate One Month After Discharge From Emergency Department for Asthmatic Patients Given a Strict Formalized Follow up Protocol
Acronym: ASUR-R
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P130943; IDRCB : 2014-A01006-41 (Other: IDRCB)
Record Dates: First submitted 2015-04-20; First posted 2015-04-23 (Estimated); Last update posted 2022-03-24 (Actual); Status verified 2022-02

CONDITIONS: Asthma
Keywords: Asthma; Relapse; Therapeutic counselling; Protocol of care
MeSH Terms: conditions — Asthma; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1: Control (Active Comparator)
  Interventions: Behavioral: 1: Control
- 2: Intervention (Experimental)
  Interventions: Behavioral: 2: Intervention

INTERVENTIONS:
Behavioral: 2: Intervention — 1. The corticoid treatment (Prednisolone or Prednisone) given from the ED for the first day if the patient is discharged at nighttime or during the weekend.
     A detailed prescription including 1) A written prescription of the corticosteroid treatment given orally for a total treatment length of 7 days 2) A written prescription describing the adaptation of the inhaled treatment 3) Peak expiratory flowmeter
  2. A written action plan with formalized recommendations for the patient
  3. A formal letter and recommendations to the general practitioner including information about the ED visit, and the necessity to program a follow up with regular consultations as well as to program spirometry evaluation for his patient.
     The ED doctor at discharge will explain all these documents orally
  4. Recommendations for an early contact with the general practitioner;
  5. Telephone call of the emergency department to the patient at day 7 +/-1 in order to ensure the link with the general practitioner.
  Arms: 2: Intervention
Behavioral: 1: Control — patients without discharge protocol
  Arms: 1: Control

SUMMARY:
For over ten years, the French group ASUR (ASthme aux URgences) has studied the asthmatic disease. The first epidemiological study enrolling 3.772 patients, in 39 emergency services, showed that the treatment protocols during the acute asthma attacks were not homogeneous and that oral corticosteroids were prescribed in only 50% of the cases. The second major French study in the emergency department by the same group enrolled 3.049 patients. The results showed that 38% of patients have a new acute asthma relapse in the month following their consultation in the emergency department. In the same study, a multivariate analysis of predictors of relapse showed that there are controllable factors (absence of written recommendations at discharge, only 50% of prescriptions for oral corticosteroids at discharge from the emergency department, limited follow-up by a general practitioner (GP) or pneumologist ...).

The emergency physician has a responsibility in educating the patient during the period between an acute asthma attack and return to the stability of long term therapy. To date, the impact of patient education on the rate of further consultations in the emergency department has not been proven, although it seems to be a positive trend on its effect. In France, half of the patients coming to the emergency department for asthma attack will not be hospitalized. More than a third will return to the ED within the first 30 days for a new attack. The impact of post-interventional education on relapse should be explored. A first major study on a strict formalized protocol designed to reduce the relapse rate is essential and could allow a major improvement.

Our main objective is to assess the impact of a strict formalized protocol of care of asthmatic patients discharged from the Emergency Department on the recurrence rate of asthma attacks, one month after an asthma attack.

The expected benefit for the patient is the short-term reduction of relapse after asthma exacerbations, thus avoiding the problems of readmission. The strict formalized discharge protocol would also improve education in terms of self-medication in this gray zone of post-therapeutic monitoring. The benefit is even more important in terms of public health due to the important prevalence of asthma in the world and in our country. The advantage of this protocol is to strengthen the links between the hospital and the GPs. Education of asthmatic patients is essential in reducing morbidity. Thus, the potential benefits of this protocol are: reducing the cost of health and re-hospitalization, improved education of asthma patients, strengthening their link with the required GP, decreased absenteeism usually frequent in this type of disease in the workplace.

DETAILED DESCRIPTION:
Main objective

To assess the impact of a strict formalized protocol of care of asthmatic patients discharged from the Emergency Department on the recurrence rate of asthma attacks, one month after an asthma attack.

Secondary objectives

Assess the impact of a strict formalized protocol on the rate of hospitalization one month after discharge from the ED.

Assess the rate of early recurrence of asthma attacks within the first 15 days after discharge from the ED.

Assess the control of the asthmatic disease at one month after discharge from the ED, by using a recognized tool, the Asthma Control Test (ACT).

Assess the compliance rate of the patients to the recommended therapeutic strategy.

Primary end point:

Recurrence rate of any asthma attacks diagnosed by the GP or the ED doctor, one month after discharge from the ED.

Secondary end points:

Recurrence rate of asthma attacks at 15 days +/-2 after discharge from the ED. Rate of hospitalization within 30 days +/-2 after discharge from the ED Score to the asthma control test (ACT) 30 days +/-2 after discharge from the ED.

Rate of patient's adherence to protocol: we will count the number of GINA (6) discharge recommendations followed in both groups Percentage of patients having purchased a peak expiratory flow meter at D30 +/-2 First day of contact with the general practitioner after leaving the Emergency Department.

Percentage of patients' follow-up by the general practitioner at D30 +/-2 Percentage of patients using their peak expiratory flow meter at D30 +/-2. We will classify four categories of use of PEF: daily, weekly, less than once a week, never.

Percentage of patients self-medicating before calling the doctor Experimental plan Multicenter, prospective, cluster-randomized, open study, enrolling a cohort of patients who were managed in the emergency department for an acute asthma attack and who have no admission criteria at the end of treatment. Forty-six Emergency Departments will be selected on the national territory, randomized by cluster (centers A [control=standard group], centers B [treatment group= strict formalized protocol] and stratified by size (number of patients per year) and types [CHU, CHG, CHR]).

The two groups of patients will be contacted by telephone at Day 15 +/-2, and Day 30 +/-2 of discharge in order to identify a possible relapse, to collect the various elements of the evolution of their disease as well as a to answer a formalized questionnaire.

Relapse is defined as a respiratory discomfort due to asthma and requiring medical assistance (in the emergency department or with the GP).

Number of patients needed: A sample size of N= 466 patients/group allow 80% power to detect a 30% relative difference in recurrences (i.e. from 25% to 17.5%) with a chi-square test and a two-sided 5% significance level. Considering an attrition rate around 5% and that the study is a cluster- randomized design, we applied a variance inflation factor equal to 1.5 (based on previous studies) .

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria :

Patients over 18 years, consulting to the Emergency room for an acute asthma attack which, after initial treatment is discharged directly from the ED having given his free and informed consent, and affiliated to the social security.

Exclusion Criteria:

* Impossibility to a correct follow up (foreigners who do not live in France, language barrier, homeless, no social security).
* Wheezing of other origin:

  * Infectious pneumonia
  * Acute cardiac failure
  * COPD
* Immediate resuscitation criteria: respiratory failure or pause, RR < 10/min, and CGS <8
* PEFR<50% four hours after arrival in the ED
* Patient under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1422 (Actual)
Dates: Start 2015-08; Primary Completion 2022-02-16 (Actual); Study Completion 2022-02-16 (Actual)

PRIMARY OUTCOMES:
Recurrence rate of any asthma attacks diagnosed by the GP or the ED doctor, one month after discharge from the ED | 1 month

SECONDARY OUTCOMES:
Recurrence rate of asthma attacks at 15 days +/-2 after discharge from the ED | 2 weeks
Rate of hospitalization within 30 days +/-2 after discharge from the ED | 1 month
Score to the asthma control test (ACT) 30 days +/-2 after discharge from the ED | 1 month
Rate of patient's adherence to protocol: we will count the number of GINA (6) discharge recommendations followed in both groups | 1 month
Percentage of patients having purchased a peak expiratory flow meter at D30 +/-2 | 1 month
First day of contact with the general practitioner after leaving the Emergency Department | 7 days
Percentage of patients' follow-up by the general practitioner at D30 +/-2 | 1 month
Percentage of patients using their peak expiratory flow meter at D30 +/-2. We will classify four categories of use of PEF: daily, weekly, less than once a week, never. | 1 month
Percentage of patients self-medicating before calling the doctor | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer TRUCHOT, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Patrick PLAISANCE, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service des Urgences, Hôpital Lariboisière, Paris, France